CLINICAL TRIAL: NCT01999179
Title: Pilot Study of Post-thrombotic Syndrome & Predictors of Recurrence in Cancer Patients With Catheter-related Thrombosis
Brief Title: Post-thrombotic Syndrome & Predictors of Recurrence in Catheter-related Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Versiti Blood Health (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Lisa Baumann Kreuziger, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO21429
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Venous Thrombosis; Neoplasms
Keywords: catheter related thrombosis; upper extremity deep venous thrombosis; central venous catheters; cancer; Catheters
MeSH Terms: conditions — Venous Thrombosis; Neoplasms | interventions — Heparin; Enoxaparin; apixaban; Rivaroxaban; Dabigatran; edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- low-molecular-weight heparin or direct oral anticoagulant (Other): Enoxaparin 1 mg/kg subcutaneously every 12 hours for one month following catheter removal or alternate enoxaparin dose or interval based on anti-factor Xa testing that was obtained by clinical team.
  Apixaban, rivaroxaban, dabigatran, or edoxaban at standard dosing per FDA package insert for direct oral anticoagulants.
  Interventions: Drug: Heparin, Low-Molecular-Weight, or direct oral anticoagulants

INTERVENTIONS:
Drug: Heparin, Low-Molecular-Weight, or direct oral anticoagulants — Cancer patients will be treated with enoxaparin 1 mg/kg subcutaneously every 12 hours for one month following catheter removal or alternate enoxaparin dose or interval based on anti-factor Xa testing obtained by the clinical team or either apixaban, rivaroxaban, dabigatran, edoxaban following a catheter related blood clot
  Other Names: enoxaparin; apixaban; rivaroxaban; dabigatran; edoxaban

SUMMARY:
The goal of the pilot study is to determine if a multicenter prospective cohort study of cancer patients with blood clots associated with catheters is feasible. Cancer patients with catheter-related thrombosis treated with one month of anticoagulation will be evaluated for for post-thrombotic syndrome. Laboratory biomarkers will be evaluated as predictors of recurrent thrombosis.

DETAILED DESCRIPTION:
Participants may be referred for screening at Medical College of Wisconsin (MCW) in two possible mechanisms: participant contact study staff from information on Clinical Trials Science Institute (CTSI) FACT website or referral from treating Hematologist or Oncologist. At MCW, an EPIC report will be generated to identify people with catheter related thrombosis (CRT). The treating provider would then be contacted to determine if referral to the study was appropriate. Subjects at Ohio State University (OSU) will be referred from the treating Hematologist or Oncologist. A report generated in Epic will be used to identify people with CRT. The treating provider would then be contacted to determine if referral to the study was appropriate. Participants will be given printed information about the study or verbal explanation using the informational flyer. Verbal consent will be obtained to be screened for participation and contacted by study personnel. Screening will be completed by BloodCenter of Wisconsin (BCW) nurse coordinator. We aim to consent and enroll patients after diagnosis of catheter-related thrombosis and prior to catheter removal. Consent and enrollment (Visit 1) must occur prior to discontinuation of anticoagulation. Participants will be treated with either enoxaparin for one month following catheter removal, or direct oral anticoagulant treatment (apixaban, rivaroxaban, dabigatran, or edoxaban). Anticoagulation will be continued for 1 month after catheter removal. The minimum duration of anticoagulation will be one month and maximum duration is 7 months. The cost of enoxaparin will be the responsibility of the participant as use of the medication is part of routine care. Subjects will be contacted by telephone prior to discontinuation of anticoagulation to review study protocol, assess for bleeding, and see if any continuation rules apply and arrange for research visit 2 in the following 1-2 weeks. Visits 3 and 4 will occur 3 and 6 months after catheter removal, respectively. At visits 3 & 4, Medical history, cancer history, and medications will be updated. At each visit, participants will be assessed for post-thrombotic syndrome using the modified Villalta scale and functional limitation using the DASH questionnaire. At MCW, surveys will be administered by the research coordinator and/or Translational Research Unit (TRU) staff and physical examination will be completed by BCW nurse coordinator. At OSU, surveys will be administered by research coordinators and physical examination will be administered by research nurse coordinator. Laboratory samples will be obtained for MCW participants only.

ELIGIBILITY:
Inclusion Criteria:

* Upper extremity venous thrombosis associated with an indwelling catheter documented by ultrasound, CT or venography
* Current hematologic or solid tumor malignancy undergoing chemotherapy, surgery, radiation or hormonal therapy for malignancy.
* >18 years of age
* Platelet count >50,000
* Creatinine clearance >30 ml/min
* Ability to provide informed consent

Exclusion Criteria:

* Underlying medical condition or chemotherapy requiring long-term anticoagulation
* Known underlying higher risk thrombophilias including antiphospholipid antibody syndrome, antithrombin, protein C or protein S deficiencies, or homozygosity or compound heterozygosity for prothrombin G20210A or Factor V R506Q mutations.
* Inability to remove venous catheter
* Anticipated replacement of central venous catheter within 3 months
* Major bleeding or clinically relevant non-major bleeding in the preceding 60 days
* Participation in another clinical trial that requires anticoagulation
* Use of anticoagulant other than low-molecular weight heparin
* Treatment with thrombolysis
* Catheter removal >1 month prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-06; Primary Completion 2019-04-02 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Baumann Kreuziger, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - The Ohio State University, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-molecular-weight Heparin or Direct Oral Anticoagulant: Enoxaparin 1 mg/kg subcutaneously every 12 hours for one month following catheter removal or alternate enoxaparin dose or interval based on anti-factor Xa testing that was obtained by clinical team.
  Apixaban, rivaroxaban, dabigatran, or edoxaban at standard dosing per FDA package insert for direct oral anticoagulants.
  Heparin, Low-Molecular-Weight, or direct oral anticoagulants: Cancer patients will be treated with enoxaparin 1 mg/kg subcutaneously every 12 hours for one month following catheter removal or alternate enoxaparin dose or interval based on anti-factor Xa testing obtained by the clinical team or either apixaban, rivaroxaban, dabigatran, edoxaban following a catheter related blood clot
Period: Overall Study
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
Started | 27
Completed | 20
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Change in Therapy | 3
Not completed — New catheter | 2

BASELINE CHARACTERISTICS:
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
Number analyzed (Participants) | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [48 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: PTS Assessment Completion
Description: Percentage of participants who completed post-thrombotic syndrome assessments
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
Number analyzed (Participants) | 27
Participants | 17

2. Secondary Outcome: Biomarker Sample Collection
Description: Number of participants that completed sample collection for biomarker analysis to predict recurrent venous thrombosis
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
Number analyzed (Participants) | 12
participants | 7

3. Other Pre Specified Outcome: Number of Participants With Post-thrombotic Syndrome
Description: The number of participants with post-thrombotic syndrome 6 months after catheter removal in cancer patients with catheter-related thrombosis treated with 1 month of anticoagulation
Time Frame: 6 months after catheter removal
Measure: Count of Participants; unit: Participants
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
Number analyzed (Participants) | 20
Participants | 0

4. Other Pre Specified Outcome: Number of Participants With Recurrent Thrombosis
Description: Number of participants with recurrent thrombosis in cancer patients with catheter-related thrombosis treated with 1 month of anticoagulation
Time Frame: 6 months after catheter removal
Measure: Count of Participants; unit: Participants
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
Number analyzed (Participants) | 20
Participants | 0

5. Other Pre Specified Outcome: Number of Participants With Major Bleeding
Description: Number of participants with major bleeding in cancer patients with catheter-related thrombosis treated with 1 month of anticoagulation
Time Frame: 6 months after catheter removal
Measure: Count of Participants; unit: Participants
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
Number analyzed (Participants) | 20
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Low-molecular-weight Heparin or Direct Oral Anticoagulant
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27
Other Adverse Events (participants affected / at risk) | 2/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-molecular-weight Heparin or Direct Oral Anticoagulant (N=27)
Hematoma (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low-molecular-weight Heparin or Direct Oral Anticoagulant (N=27)
Bleeding (Blood and lymphatic system disorders) | 2
Fall (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT01999179/Prot_SAP_000.pdf